CLINICAL TRIAL: NCT05803902
Title: A Randomized, Double-blind, Dose-escalation Phase I Clinical Study to Evaluate the Safety, Tolerability and Pharmacokinetics of 9MW1911 Injection in Healthy Subjects
Brief Title: An Evaluation of 9MW1911 Injection in Healthy Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Mabwell (Shanghai) Bioscience Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 9MW1911-2021-CP101
Record Dates: First submitted 2022-03-29; First posted 2023-04-07 (Actual); Last update posted 2025-12-15 (Actual); Status verified 2025-12

CONDITIONS: Asthma; COPD; Atopic Dermatitis
MeSH Terms: conditions — Asthma; Pulmonary Disease, Chronic Obstructive; Dermatitis, Atopic

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (8):
- 9MW1911 Dose 1 (Experimental): 9MW1911 injection ( Dose 1) by intravenous injection once on the first day of treatment. 8 subjects will be enrolled, including 2 subjects for placebo administration.
  Interventions: Drug: Experimental drug 9MW1911; Drug: Placebo
- 9MW1911 Dose 2 (Experimental): 9MW1911 injection (Dose 2) by intravenous injection once on the first day of treatment. 8 subjects will be enrolled, including 2 subjects for placebo administration.
  Interventions: Drug: Experimental drug 9MW1911; Drug: Placebo
- 9MW1911 Dose 3 (Experimental): 9MW1911 injection (Dose 3) by intravenous injection once on the first day of treatment. 8 subjects will be enrolled, including 2 subjects for placebo administration.
  Interventions: Drug: Experimental drug 9MW1911; Drug: Placebo
- 9MW1911 Dose 4 (Experimental): 9MW1911 injection (Dose 4) by intravenous injection once on the first day of treatment. 8 subjects will be enrolled, including 2 subjects for placebo administration.
  Interventions: Drug: Experimental drug 9MW1911; Drug: Placebo
- 9MW1911 Dose 5 (Experimental): 9MW1911 injection (Dose 5) by intravenous injection once on the first day of treatment. 8 subjects will be enrolled, including 2 subjects for placebo administration.
  Interventions: Drug: Experimental drug 9MW1911; Drug: Placebo
- 9MW1911 Dose 6 (Experimental): 9MW1911 injection (Dose 6) by intravenous injection once on the first day of treatment. 8 subjects will be enrolled, including 2 subjects for placebo administration.
  Interventions: Drug: Experimental drug 9MW1911; Drug: Placebo
- 9MW1911 Dose 7 (Experimental): 9MW1911 injection (Dose 7) by intravenous injection once on the first day of treatment. 8 subjects will be enrolled, including 2 subjects for placebo administration.
  Interventions: Drug: Experimental drug 9MW1911; Drug: Placebo
- 9MW1911 Dose 8 (Experimental): 9MW1911 injection (Dose 8) by intravenous injection once on the first day of treatment. 8 subjects will be enrolled, including 2 subjects for placebo administration.
  Interventions: Drug: Experimental drug 9MW1911; Drug: Placebo

INTERVENTIONS:
Drug: Experimental drug 9MW1911 — Experimental drug administered with IV infusion
Drug: Placebo — Placebo administered with IV infusion

SUMMARY:
This study is a randomized, double-blind, dose-escalating phase I clinical study to evaluate the safety, tolerability and pharmacokinetics of 9MW1911 injection in healthy subjects.

ELIGIBILITY:
Inclusion Criteria:

- 1. Male or female subjects aged 18 to 65 years (including 18 and 65 years). 2. Weight≥50.0 kg for males, or weight≥45.0 kg for females, and body mass index (BMI) in the range of 19.0 ~ 26.0 kg/m2 (including cut-off value).

3. Female subjects must have a negative β-HCG pregnancy test (Screening and Baseline); Subjects(including their partners) will take effective contraceptive measures voluntarily.

Exclusion Criteria:

* 1. Subjects who have a history of allergies to biological agents or any drug components; those who have a history of allergies and judged by the investigator to be ineligible for enrollment.

  2. The clinical laboratory tests show any clinical abnormalities, or abnormalities with clinical significance (including but not limited to diseases of digestive tract, kidney, liver, nervous system, blood, endocrine system, cancer, lung, immune system, mental, heart) , and judged by the investigator to affect participation in this study.

  3. Subjects with prolonged QTcF interval (> 450 ms) on electrocardiogram (ECG) examination, or family history of prolonged QTc syndrome or sudden death.

  4. Subjects received any biological treatment (including all vaccines except the coronavirus vaccine) within 3 months before screening, or planned to take biological treatment during the study period, or received the new coronavirus vaccine within 1 month before screening.

  5. Subjects received any prescription drugs or traditional Chinese medicines, including vitamins, trace elements or dietary supplements within 14 days before screening; except for topical products without systemic absorption.

  6. Subjects with a history of smoking within 6 months before screening, or unwilling to stop smoking during the study, or willing to use products containing nicotine during the study.

  7. Subjects who have lost blood or donated blood ≥200mL within 3 months before screening, or those who plan to donate blood within 3 months.

  8. Subjects positive screening for viral hepatitis (including hepatitis B and C), HIV antibodies, and Treponema pallidum antibodies.

  9. Subjects who paticipated any clinical trial within 3 months before screening.

  10. Subjects who is inappropriate to participate in the trial due to any reasons as determined by the investigator.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 48 (Actual)
Dates: Start 2021-12-15 (Actual); Primary Completion 2023-03-06 (Actual); Study Completion 2023-03-06 (Actual)

PRIMARY OUTCOMES:
Adverse Event(including serious adverse event) | Day0-Day113
  Evaluate the safety and tolerability of 9MW1911 in healthy subjects, and to determine the possible maximum tolerated dose (MTD).

SECONDARY OUTCOMES:
Pharmacokinetics parameters | Day0-Day113
  Maximum concentration(Cmax)
Pharmacokinetics parameters | Day0-Day113
  The area under the curve (AUC)
Pharmacokinetics parameters | Day0-Day113
  Time at which maximum concentration(Tmax)
Pharmacokinetics parameters | Day0-Day113
  The half life(T1/2)
Immunogenicity parameters | Day0-Day113
  The incidence of ADAs against 9MW1911 during the study will be summarized

CONTACTS AND LOCATIONS:
Locations (1):
- Peking Union Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided